CLINICAL TRIAL: NCT05614830
Title: Effectiveness of Dry Needling in Management of Myofacial Trigger Point In Trapezius Muscle
Brief Title: Effectiveness Taif University P. O. Box 11099 Taif 21944 Effectiveness of Dry Needling in Management of Myofacial Trigger Point
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Slwa Sami Alattar, Student, Taif University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44-004
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Myofacial Trigger Points
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Dry needling ,
- Control group (Active Comparator): Usual physical therapy protocol 4 sessions, two sessions per week each session will include a group of therapeutic exercises
  Interventions: Other: usual physical therapy program

INTERVENTIONS:
Other: Dry needling , — The intervention group will receive sessions of dry needling to relief myofacial pain on trapezius
  Arms: Intervention group
Other: usual physical therapy program — Therapeutic exercise
  Arms: Control group

SUMMARY:
myofascial pain syndrome is considered to be a chronic condition due to sensitive pressure points within the muscle recognized as trigger points

Generally the aim of this study will be :

* To investigate the effectiveness of dry needling on trigger point in trapezius muscle
* Evaluate the pain level before and after the applications of dry needling on trigger points
* compare between the effects of dry needling and physical therapy exercise program

ELIGIBILITY:
Inclusion Criteria:

* Clinically active trigger point and expression of symptoms of neck pain in trapezius which had lasted for at least 3 months.
* Having a pain level higher than 4 and lower than 8 on Visual Analogue Scale ( VAS )
* Did not receive any other form of neck treatment during the previous month.

Exclusion Criteria:

* Presence of cardiopulmonary disease , the application process requires the subject to be in prone position to expose the area of treatment, this position is un-preferable for cardiopulmonary patients
* History of neck surgery
* Trigger point treatment in the last 30 days
* Any contraindications for dry needling such as local infection, skin disease ,severe postural disorder , tumor , rheumatoid arthritis, cervical spine stenosis and bilateral upper extremity symptoms
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Pain level | 6 weeks
  Will be determined using the visuals analogue scale (VAS)
Neck disability index | 6 weeks
  questionnaire contains 10 items aiming to evaluate the limitation because of neck pain

SECONDARY OUTCOMES:
Depression | 6 weeks
  Will be determined using the Beck's Depression Inventory ( BDI)
Neck Range of motion | 6 weeks
  Will be measured using CROM